CLINICAL TRIAL: NCT02854735
Title: Non-invasive Total Body Composition in Early Detection of Nutrition Depletion, Changes in Body Physiology and Treatment Response in Head and Neck Patients Undergoing Concurrent Chemoradiotherapy
Brief Title: Total Body Composition in Detection of Nutrition Depletion in Head and Neck Patients
Acronym: TBCHNC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMRPG2E0101
Record Dates: First submitted 2016-08-01; First posted 2016-08-03 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-07

CONDITIONS: Head and Neck Neoplasms; Dual-Energy X-Ray Absorptiometry; Malnutrition
Keywords: Head and Neck Neoplasms; Total body composition; Dual-Energy X-Ray Absorptiometry; Malnutrition; Muscle quantification
MeSH Terms: conditions — Head and Neck Neoplasms; Malnutrition | interventions — Densitometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Head and neck neoplasm: Patients with stage III-IV head and neck cancer (squamous cell carcinoma) patient undergoing CCRT
  Interventions: Other: Imaging by CT and densitometry

INTERVENTIONS:
Other: Imaging by CT and densitometry — Imaging by CT and densitometry, no intervention involved

SUMMARY:
The purpose of this study is to define the role of total body composition in the guidance of nutritional support and treatment monitoring in head and neck patients. Furthermore, the second aim of this study is to compare the clinical performance of dual energy X-ray absorptiometry as compared to CT in evaluating total body composition of patients.

DETAILED DESCRIPTION:
In this 4-year cohort study, a total of 120 patients with stage III-IV head and neck cancer (squamous cell carcinoma) patient undergoing concurrent chemo-radiotherapy will be enrolled. Laboratory examination will be performed to evaluate the physiological change and treatment related toxicity, including BUN and Cr for hydration and renal function; complete blood cell and differential count, pre-albumin and albumin for nutrition, and C-reactive protein for inflammatory change. Both CT and dual energy X-ray absorptiometry (DXA) will be used to evaluate total body composition. CT is used to evaluate surface area of fat and muscle, and DXA is used to evaluate lean body mass, fat body mass and bone mineral content. MRI of the head and neck region is used for tumor staging of the head and neck cancer, monitoring the treatment response and detecting treatment related adverse effect.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven head and neck (SCC), surgery of the primary tumor/lymph nodes is limited to incisional/excisional biopsy.
2. 2010 7th edition AJCC stage III, IVA (T4N0-2) and IVB (any T, N3).
3. Well-informed and accepted treatment of CCRT.
4. Age 20-70 years old.
5. Negative pregnancy test for women of childbearing potential.
6. Adequate hematopoietic or organ function which is amenable for chemotherapy:

   * A leukocyte count ≥3000/L
   * Platelet count ≥100,000/L.
   * Serum bilirubin level ≦ 1.5mg/dL
   * Serum creatinine level ≦1.6 mg/dL or creatinine clearance ≥ 60 mL/min/1.73 m2.
   * ALT/AST ≦ 3X ULN

9. Ability to understand and willingness to be enrolled in our study and sign a written informed consent document

Exclusion Criteria:

1. NPC is excluded from this study.
2. Patients have acute medical conditions (such as bacterial or viral infection or active cardiopulmonary disease) that may be incapable of having regular image study.
3. Patients are under regular steroid or hyperthyroid medications, which may have great impact on the whole body metabolism.
4. Patients are under-nutrient and they need to have regular liquid oral nutrition formulas support.
5. Patient that have dementia or pregnant.
6. Patients not expecting to comply with follow up.
7. Patient not suitable for chemotherapy.
8. Patient not suitable for MRI, such as claustrophobia, previous metal implantation, previous cardiac pacemaker implantation, inability to comply with MRI instructions and poor renal function.
9. Received barium study within a week.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage III-IV head and neck cancer (squamous cell carcinoma) patient undergoing concurrent chemo-radiotherapy for cancer treatment
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Alterations of the total body composition | 3 years
  Determine the alterations of total body composition in response to physiological change during the course of the cancer treatment, thus allowing clinicians to understand the optimal time for administering additional nutritional support during the CCRT treatment.

SECONDARY OUTCOMES:
Comparison of densitometry with CT | 3 years
  To compare the performance of densitometry to CT in the evaluation of total body composition as a marker for monitoring cancer treatment related changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Guishan, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Depending on IRB regulation